CLINICAL TRIAL: NCT04628234
Title: Follow-up of Actual Patient Care Site Two Months After Hospitalisation Compared With Their Expressed Choice Regarding Subsequent Care Site
Brief Title: Follow-up of Actual Patient Care Site Two Months After Hospitalisation Compared With Their Expressed Choice Regarding Subsequent Care Site (RESPECT)
Acronym: RESPECT
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-001; 2020-A00439-30 (Other: IDRCB)
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hematologic Malignancy; Tumor, Solid
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an onco-hematologic solid tumor in palliative care

SUMMARY:
This is a non randomized, monocentric, descriptive, transversal and prospective study. The purpose of this study is to assess the compliance with patient expressed choice regarding subsequent care and death -if occured- site (at hospital or at home) after hospitalisation for terminally ill patients with an onco-hematologic solid tumor in palliative care and to identify reasons for potential non-compliance.

DETAILED DESCRIPTION:
Patients will reply to two questionnaires, at inclusion and two months after inclusion. Primary care physician will also be contacted by phone to reply to two questionnaires, at inclusion and two months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old
* Patients with onco-hematologic solid tumor (locally advanced or metastatic) against which specific and systemic treatments are outdated or have been stopped (symptomatic palliation with radiotherapy is allowed)
* Patients admitted in full hospitalisation
* Patients able to speak, read and understand French
* Patients able to answer the phone
* Signed informed consent from the patient
* Patients must have a social security coverage

Exclusion Criteria:

* Patients < 18 years old or incapable person ≥ 18 years old
* Patients admitted for any surgical intervention
* Patients unable to read French
* Patients whose physical or psychological condition do not allow them to answer orally or in writing
* Patients deprived of liberty
* Patients placed under judicial protection
* Women that are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an onco-hematologic solid tumor in palliative care
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2020-07-04 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Number of patients for which their choice of care and death -if occured- site (at hospital or at home) is respected. | 2 months after inclusion
  Patients will fill out a questionnaire at inclusion and 2 months after inclusion if they are still alive. Death site will be collected from primary care physician if patient died.
  The patient expressed choice regarding subsequent care and death site collected in the first questionnaire at inclusion will be compared to the situation at 2 months.

SECONDARY OUTCOMES:
Number of new hospitalisations occuring after inclusion, if any. | 2 months after inclusion
Duration of new hospitalisations occuring after inclusion, if any. | 2 months after inclusion
Reasons for new hospitalisations occuring after inclusion, if any. | 2 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Cancerologie Strasbourg Europe, Strasbourg, France